| 1 | RinasciMENTE. An Internet-Based Self-Help Intervention to Cope with Psychological Distress |
|---|---|
| 2 | Due to COVID-19: A Study Protocol for a Randomized Controlled Trial |
| 3 | |
| 4 | |
| 5 | NCT04907903 |
| 6 | |
| 7 | Version: 02/02/2022 |
| 8 | |
| 9 | |
| 10 | |
| 11 | |
| 12 | |
| 13 | |
| 14 | |
| 15 | |
| 16 | |
| 17 | |
| 18 | |
| 19 | |
| 20 | |
| 21 | |
| 22 | |
| 23 | |
| 24 | |
| 25 | |
| 26 | |

## **ABSTRACT**

27

28 **Background** This study aims to evaluate the feasibility and effectiveness of the RinasciMENTE 29 program, an Internet-based self-help intervention based on Cognitive Behavioral Therapy (CBT) 30 principles and techniques in supporting individuals experiencing psychological impairments during 31 the COVID-19 pandemic. A randomized controlled trial (RCT) design with random allocation at the 32 level of individual will be conducted to compare the impact of the RinasciMENTE program with a 33 waiting list control in improving the psychological functioning of the general population during the 34 COVID-19 pandemic. Methods A minimum sample of 128 participants experiencing mild/subthreshold levels of 35 36 psychological symptoms during the COVID-19 pandemic will be recruited. After the initial 37 screening, participants will be randomly assigned to either the experimental group or the control 38 condition. The program will last 2 months, during which participants will receive 8 weekly CBT 39 treatment modules. The impact of the RinasciMENTE program on selected primary and secondary 40 psychological outcomes will be tested at the end of the intervention (2 months), 6- and 12-month 41 follow-up. 42 **Discussion** We expect people to show an increased level of psychological functioning, and to acquire the skills and self-confidence necessary to deal with the psychological consequences of the COVID-43 44 19 outbreak and its related social isolation during and following the pandemic. 45 Trial registration ClinicalTrials.gov NCT0497903 Registered on 28 May 2021.

46

- 47 Keywords: COVID-19, Internet-based intervention, Self-help, Cognitive-behavioral therapy,
- 48 Psychological distress, Randomized controlled trial, Clinical psychology.

49

50

51

### **BACKGROUND**

53

54 In the hope of reducing the transmission of Coronavirus Disease 2019 (COVID-19) governments around the world have implemented unprecedentedly strict preventive measures, such as home 55 56 confinement, mobility restrictions, and social distancing (1, 2). However, the COVID-19 pandemic 57 and the resulting economic recession (3) have negatively affected the mental health of many people 58 (4). The most common mental disorders emerging were anxiety and depression, obsessive-59 compulsive symptoms, insomnia, and post-traumatic stress disorder symptoms (5-9). These were not 60 only a direct consequence of the pandemic but also largely driven by the effects of prolonged social isolation. Although necessary to limit the spread of the epidemic, social isolation resulted in increased 61 62 sedentary lifestyle (2) and other COVID-19-related stressors including fears of infection, frustration 63 and boredom, and lack of in-person contacts (10, 11). Italy was one of the most affected countries 64 during the outbreak, initially accounting for over 223.000 infected individuals and more than 31.000 65 deaths (12). In May 2021, 4.111.110 people resulted having contracted the virus, and 122.833 of them 66 died as a consequence (13, 14). 67 In this scenario, it is crucial to assess the level of psychological distress and to provide ad hoc 68 psychological interventions to support the individuals' wellbeing in both the general population (15, 69 16) and at-risk groups (17, 18) during the COVID-19 pandemic. 70 Accordingly, evidence from previous epidemics highlights the risk for long-term mental health issues 71 (19) and emphasizes the need for continued support during and after the pandemic (20). 72 Many health organizations have already committed resources to support the mental well-being of the 73 individuals, adapting existing standard programs to meet evolving demands caused by COVID-19 74 (21). In this regard, cognitive-behavioral techniques including restructuring of cognitive bias, as well as activity planning and relaxation, have been shown particularly useful in addressing psychological 75 76 distress (22-25).

77 Cognitive-behavioral therapy (CBT) is a time-sensitive, structured, present-oriented psychotherapy 78 aimed at helping people identify and change thinking and behavior patterns that are harmful or 79 ineffective, replacing them with more accurate thoughts and functional behaviors. 80 Still, given that face-to-face treatment is not always viable in these circumstances (26) a new way to 81 deliver psychological treatments is urgently required, and a potentially practical solution is to deliver 82 therapy remotely (14, 27-30). 83 Many systematic reviews and randomized controlled trials (RCTs) demonstrated the utility and the 84 efficacy of Internet-based interventions in supporting people experiencing psychological problems 85 (31-33).86 Advantages include improved access for individuals (26) who have variable schedules, an important 87 workload, or who are afraid of being contaminated through face-to-face contacts (34-36), as well as 88 cost-effectiveness compared to face-to-face treatment. 89 Due to its features, CBT well-suits many aspects of distance therapy. First, it is a talking therapy, and 90 this aspect can be relatively easily retained remotely. It also emphasizes the importance of the person 91 making changes and working on specific tasks between sessions to bring about the change (37); this 92 is perfectly consistent with working remotely. Moreover, with distance therapy, the patient may be 93 less likely to attribute the progress to the therapist and more likely to have an improved sense of self-94 efficacy (38). One of the goals of CBT is to "become your therapist" by learning skills people can use 95 on their own after treatment to keep feeling well. 96 Research shows that CBT delivered digitally (iCBT) is effective in reducing symptoms of social 97 anxiety disorder (39, 40), generalized anxiety disorder (41, 42), panic disorder (43), major depressive 98 disorder (44-46), obsessive-compulsive disorder (47) and insomnia (48) in both guided and unguided 99 self-help programs. Specifically, a review of 30 studies found that CBT-based self-help interventions 100 significantly reduced both anxiety and depression. Studies also show that people tend to maintain 101 their progress over time, which is very encouraging (49). Furthermore, since patients can return to

102 the program at their convenience to access treatment information, this may facilitate learning and 103 retention. 104 Despite a growing interest in the field of web-based psychological interventions, Internet-based CBT 105 self-help programs remain underdeveloped. 106 To fill this important gap in the literature and to properly meet the need of the population, it is crucial to promote and investigate the impact of this Internet-based psychological intervention in increasing 107 108 individuals' emotional well-being. 109 For this reason, the present RCT aims to explore the effectiveness of a novel Internet-based CBT self-110 help program specifically developed to address the immediate stress and prevent long-term 111 psychological consequences of the COVID-19 pandemic among Italians both living in the county and 112 abroad. To assess its impact, the effects of the RinasciMENTE program will be compared with a waiting list (WL) condition on selected self-reported measures immediately following the 8-week 113 114 intervention and at 6- and 12-month follow-up. 115 The primary hypothesis that will be tested is that the program will be feasible and effective in 116 increasing the psychological functioning of the person. 117 The secondary hypothesis will test whether participants assigned to the experimental condition will 118 show a reduced level of stress, anxiety, depression, and fear of COVID-19, as well as improved 119 emotion regulation strategies, self-efficacy, and psychological well-being than those in the WL 120 condition at treatment termination. 121 Moreover, participants in the experimental condition will be expected to present maintained outcomes 122 or further decreased psychological symptoms at 6 and 12-month after the end of the treatment 123 program.

## **METHODS**

## 125 **Design**

- The project consists of a prospective, randomized, open, and parallel group-controlled study with two
- arms: an experimental arm with 8 online weekly CBT self-help sessions, and a waiting list (WL)
- 128 control arm.

134

## 129 Ethical Statement

- The study was approved by the Ethical Committee of the Catholic University of Milan, Italy (ID: 25-
- 131 21). All procedures performed in the study will be run following the ethical standards of the
- institutional and/or national research committee and with the Helsinki Declaration and its later
- amendments or comparable ethical standards.

## Patients and public involvement

- Participants from the general population will be recruited through advertisements placed on social
- media platforms (i.e., Facebook, Instagram, Twitter), and online webinars on the topic.
- 137 The recruitment materials will include details about the study aim, the treatment delivered, and the
- conditions for participation, together with the weblink to access the program.
- 139 Inclusion criteria for the participants into the study will be: (A) being fluent in the Italian language;
- 140 (B) being over 18 years old; (C) providing online informed consent; and (D) showing
- mild/subthreshold levels of symptoms at the 12-Item General Health Questionnaire (GHQ-12) -
- 142 Italian version (50, 51) the most extensively used screening tool assessing the severity of common
- mental disorders over the past few weeks using a 4-point Likert-type scale (from 0 to 3). Its total
- score ranges from 0 to 36, with high scores indicating worse health status. Only participants who
- score  $\geq$  15 on the GHQ and show moderate levels of symptoms at the clinical interview will be
- included in the study.
- Participants will be excluded from the program if: (A) presenting visual, hearing, or cognitive
- impairments that will prevent them from receiving and following the intervention; (B) suffering from
- severe psychiatric disorders according to the Diagnostic and Statistical Manual of Mental Disorders
- 150 (DSM 5) (52); (C) lacking basic computer skills or internet access.

Respondents will not be excluded if already receiving psychopharmacological therapy or psychological-psychotherapeutic support.

# Sample size calculation

The minimum sample size required to conduct this study was calculated using an a priori sample size calculator (G\*Power 3.1.9.2 software) for F tests (53-55). Participants were randomly divided into two groups: (A) iCBT self-help and (B) waiting list control. Moreover, participants will be measured in 3 moments: (1) before the intervention, (2) at the end of intervention (two months later), and (3) after 12 months from treatment termination. Due to the novelty of the study from which to derive realistic estimates of effect sizes, the partial  $\eta$ 2 was set a priori to assume a value of 0.02 – small effect size (56, 57) – which provides a Cohen's f value of 0.143. Moreover, the type I error ( $\alpha$ ) rate was set at 0.05 (two-sided) and the Power (1 –  $\beta$ ) was set at 0.95, and the a priori correlation between repeated measures was set at 0.50, according to general guidelines (56). Lastly, the non-sphericity correction was set to 1. Results showed that there is a 95% chance of correctly rejecting the null hypothesis of no significant effect of the interaction with 128 participants in total (64 for each group).

## Randomization and blinding

The random randomization scheme will be generated using the Web site Randomization.com (58). Allocation concealment will be ensured by the program generating an anonymous code for each participant that will be associated with the randomization sequence. Due to the nature of the intervention, the treatment group allocation cannot be concealed from the participants, nor the research team and assessor of outcomes. Participants will be assigned to one of two conditions within 2 working days from their baseline assessment (Figure 1).

\*\*\* PLEASE INSERT Figure 1: Flow chart of the RinasciMENTE study

# Measures

Demographic and clinical information. Information about age, gender, education, civil status, weight, and high - used to calculate the Body Mass Index (BMI, kg/m²) in presence of dysfunctional eating behaviors - will be self-reported online at baseline. Subjects will be also asked to provide information about the country where they are currently living, their work situation (before and after the COVID-19 pandemic), and the personal experience they made of both COVID-19 pandemic and related preventive measures. The Italian version of the following psychological measures will be also collected at baseline (T0), treatment termination after 2 months (T1), at 6-month (T2), and 12-month (T3) follow-up in the experimental condition only). Please see Figure 2 for a detailed project timeline.

# \*\*\* INSERT GANTT Figure 2: Gantt of the RinasciMENTE study

Primary outcome:

175

176

177

178

179

180

181

182

183

- Outcome Questionnaire (OQ-45) (59) composed by 45 items rated on a 5-point Likert scale (0 = Never –
- 186 4 = Almost always) assessing the treatment progresses across 3 different domains: Symptom Distress (SD
- 187 25 items: 2, 3, 5, 6, 8, 9, 10, 11, 13, 15, 22, 23, 24, 25, 27, 29, 31, 33, 34, 35, 36, 40, 41, 42 and 45),
- 188 Interpersonal Relations (IR 11 items: 1, 7, 16, 17, 18, 19, 20, 26, 30, 37 and 43), and Social Role (SR –
- 9 items: 4, 12, 14, 21, 28, 32, 38, 39 and 44). The OQ-45 total score is calculated by summing the score of
- the three subscales. Total score (range 0 to 180) is calculated by the sum of the items.
- 191 Secondary outcomes:
- 192 Perceived stress scale (PSS) (60), composed of 10 items rated on a 5-point Likert scale (from 0 = never to
- 193 4 = very often) assessing the degree to which situations in one's life are appraised as stressful. PSS scores
- are obtained by reversing responses (i.e., 0 = 4, 1 = 3, 2 = 2, 3 = 1 and 4 = 0) to the four positively stated
- items (items 4, 5, 7, and 8) and then summing across all scale items. The total score (range 0 to 40) is
- calculated by the sum of the items.
- 197 Emotional regulation questionnaire (ERQ) (61), composed of 10 items rated on a 7-point Likert scale
- 198 (from 1 = strongly disagree to 7 = strongly agree) assessing respondents' tendency to regulate their

- emotions in two ways: Cognitive Reappraisal (items 1, 3, 5, 7, 8, and 10) and Expressive Suppression (items 2, 4, 6, and 9). The total score (range 7 to 70) is calculated by the sum of the items.
- Depression Anxiety Stress Scales-Short Version (DASS-21) (62), composed by 21 statements rated on a 201 202 4-point Likert scale (from 0 = did not apply to me at all to 3 = applied to me very much) assessing the 203 negative emotional states of depression, anxiety, and stress. Each of the three DASS-21 scales contains 7 204 items: Depression: dysphoria, hopelessness, devaluation of life, self-deprecation, lack of 205 interest/involvement, anhedonia, and inertia - (Items 3, 5, 10, 13, 16, 17, and 21); Anxiety: autonomic 206 arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect -(Items 2, 4, 7, 9, 15, 19, and 20); Stress: levels of chronic nonspecific arousal, difficulty relaxing, 207 208 nervous arousal, and being easily upset/agitated, irritable/over-reactive and impatient - (Items 1, 6, 8, 209 11, 12, 14, and 18). Sum scores are computed by adding up the scores on the items per (sub)scale and 210 multiplying them by 2. Sum scores for the total DASS-total scale thus range between 0 and 126, and 211 those for each of the subscales may range between 0 and 42. Ranges of scores correspond to levels 212 of symptoms, ranging from "normal" to "extremely serious". Notably, the DASS-21 has been recently 213 used to investigate the impact of the COVID-19 pandemic on the physical and mental health of 214 different populations worldwide (63-65).
- Fear of COVID-19 Scale (FCV-19S) (66) composed by 7-item rated on a 5-point scale, ranging from 1

  (from 1 = strongly disagree to 5 = strongly agree) reflecting cognitive, emotional, behavioral, and physiological manifestations of fear related to COVID-19. The total score (range 7 to 35) is calculated by the sum of the items. All items are positively worded, implying that higher scores indicate greater levels of fear.
- General Self-efficacy Scale (GSES) (67), composed of 10 items rated on a 4-point Likert scale (from 1 = Not at all true to 4 = exactly true) assessing the individuals' confidence in their ability to cope with a variety of difficult or stressing situations. The total score is calculated by finding the sum of

all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.

World Health Organization Quality of Life (WHOQOL)-BREF (68), composed of 26 items rated on a 5-point Likert scale assessing four domains: physical health (7 items on mobility, daily activities, functional capacity, energy, pain, and sleep), psychological health (6 items on self-image, negative thoughts, positive attitudes, self-esteem, mentality, learning ability, memory concentration, religion, and the mental status), social relationships (3 items on personal relationships, social support, and sex life), and environmental health (8 items related to financial resources, safety, health, and social services); it also contains QOL and general health items. The scores (range 25 to 130) are transformed linearly to a 0–100-scale.

Moreover, *adherence* will be measured through indicators such as the percentage of visited pages or the number of accesses.

Acceptability will be assessed by registering the participants' attrition rates and – for the experimental group only - by the use of the *System Usability Scale* (SUS)(69) composed of 10 statements scored on a 5-point Likert scale (from 1 = strongly disagree to 5 = strongly agree). The final score range from 0 to 100, with a score above 68 indicating the absence of usability problems.

#### **Procedure**

Those interested in taking part in the program will be directed to the RinasciMENTE website (<a href="https://www.iterapi.se/sites/rinascimente/login">https://www.iterapi.se/sites/rinascimente/login</a>) where they will find the written (online) consent, and after the acceptance of this, to each participant will be sent a document with information on the aims and requirements of the study.

They will be first asked to complete the GHQ-12 self-report questionnaires. Then, during the

following 5 days, they will choose a time slot to be contacted for a clinical semi-structured interview

248 lasting about 45 minutes, led by a certified clinical psychotherapist not involved in the study who will 249 further assess the individual's eligibility to take part in the study. Additional information about the 250 study and the randomization procedure will be also given to all respondents. 251 Next, the inclusion of each participant in the study and modules comprising the program will be 252 discussed in a group by the professional who will conduct the interview and the research investigators 253 (GP and VB), and the decision will be e-mailed to each participant within a week. Reasons for 254 exclusion will be explained to the persons and – in presence of severe psychological disturbance -255 individuals will be suggested to ask for professional help. 256 Eligible subjects will be then randomly assigned to either the experimental (iCBT self-help) or control 257 group (WL), and will receive an e-mail with a username and a customized link to create their 258 password allowing them to log into the *iterapi* platform (70, 71). The *iterapi* is a safe platform with 259 demonstrated efficacy in reducing symptoms of a wide range of disorders including somatic problems 260 - such as hearing loss (72) and tinnitus (73) - to more traditional forms of psychological suffering, 261 such as anxiety (74) and depression (75). 262 Participants in the experimental group will be required to make their first access to the platform and 263 sign an electronic informed consent form within 24 hours, while those in the control condition will 264 be able to access the online treatment once the experimental group will conclude the intervention 265 (after two months). 266 The platform will be used for communication between the mental health professionals and the participants, for the delivery of the intervention, and the quantitative assessments. 267 268 Before entering the program, participants in the study will have to complete the self-report 269 questionnaires assessing the above selected primary and secondary outcomes (T0). 270 The treatment will consist of 8 weekly modules, for a total duration of 2 months. Seven modules 271 (Introduction, Behavioral activation, Dysfunctional beliefs, Acceptance, Stress management, 272 Problem resolution and Plan of completion and maintenance) will be maintained for all participants,

while one module will be selected tailored on the specific psychological needs of each participant.

between the following: (1) *Emotional school*; (2) *Anxiety and exposition*; (3) *Constant anxiety*; (4) *Social anxiety*; (5) *Panic attack*; (6) *Sleep quality*; (7) *Perfectionism*; (8) *Relaxation*; (9) *Management*of difficult memories. The description of each module is reported in Table 1.

277

# \*\*\* INSERT Table 1: Description of the RinasciMENTE modules

279

280

281

282

283

284

285

286

288

278

For the entire duration of the intervention, every Thursday participants will receive an e-mail communicating the update of the new material on the platform. Participants who will not access the material or that will not complete the suggested tasks and exercises will receive a weekly reminder containing a brief encouraging message every Monday.

At the end of the program (after two months – T1), participants in both conditions will be asked to fill in the baseline questionnaires again. Then, the experimental group will be also assessed after 6-and 12 months from the term of the treatment (T2 and T3) (Figure 1).

# 287 Statistical analysis

- Statistical analyses were performed using SPSS software ver. 24.0 (76).
- First, preliminary analyses will be performed to test the assumptions of both univariate and multivariate normality: if (strong) violations will be detected, robust methods or data transformation
- will be applied. Dropouts will be excluded from the study.
- A missing values analysis will be run to see if the values are Missing Completely at Random (MCAR), or if there is some pattern among missing data. If there are no patterns detected, then pairwise or listwise deletion will be done to deal with missing data. However, if the missing values analysis detects a pattern, then imputation will be done.

296

297

298

The demographic characteristics will be reported as means and standard deviations for continuous variables, and frequencies and percentages for categorical variables.

299 The chi-square statistic will be used to test the association between treatment groups and socio-300 demographic and variables (i.e., age, gender, education, civil status, job), and correlation analysis 301 will be used to test the association between quantitative variables. 302 The outcomes will be compared in the two treatment conditions using an Intention-To-Treat (ITT) 303 approach. The significance level will be set at 5%. 304 A repeated-measures ANOVA will be used to determine whether there are any between and within 305 groups differences in the selected outcomes from baseline to treatment termination. Then repeated-306 measures within group ANOVA will test outcome differences over time baseline, end of treatment, 307 6- and 12-month follow-up) in the experimental group only (. Corrected effect sizes (Cohen's d) and 308 significance at 95% confidence interval (95% CI) will be calculated for both between-group and

within-group differences, while for the total effect will be calculated the Cohen's f.

# **DISCUSSION**

309

310

311 To help and mitigate the impact of the COVID-19 pandemic on selected psychological parameters, 312 the objective of this study is to evaluate the effectiveness of an Internet-based self-help intervention 313 based on CBT principles and techniques, in reducing the level of stress, anxiety, depression, and fear 314 of COVID-19, while increasing emotions self-regulation and perceived self-efficacy of Italians both 315 living in the country and abroad. . 316 The online modality was chosen due to the current multiple barriers for face-to-face psychological 317 interventions (i.e., mobility), and its largely acknowledged advantages, including greater flexibility 318 or the possibility to reach rural or low-income population (77), and Italians living outside the country 319 who look for psychological support in their language. Also, the self-help approach to therapy will be 320 employed to further improve access to treatments and empower users to strengthen their self-321 management ability, while putting less strain on therapeutic resources (78) than conventional 322 treatments do.

# **Expected results**

324

325 The results of this RCT will provide evidence for the feasibility and effectiveness of the RinasciMENTE program in supporting the emotional well-being of the persons. Specifically, people 326 327 are expected to show reduced levels of stress, anxiety, depression, and fear of COVID-19, as well as 328 improved emotion regulation strategies, and self-efficacy. They are also expected to acquire the skills 329 necessary to deal with the psychological consequences of social isolation during and after the 330 COVID-19 outbreak. 331 Still, among the weaknesses of this study, it must be anticipated possible lack of internet access and 332 digital literacy skills of some people. 333 Non-digital natives (i.e., older people) might, indeed, experience difficulties in the use of digital tools, and social isolation can pose additional challenges to their usage (i.e., chaotic home environments, 334 335 limited privacy, or unreliable internet connection) (79). 336 The use of online intervention might also prevent effective controlling of confounding variables (i.e. 337 environmental factors) that might impact treatment outcomes (80). 338 The results from this study will help to detect and address any usability problem, as Internet-based 339 interventions, due to their characteristics and format, might be a suitable and feasible solution to 340 mitigate the psychological impact of the virus outbreak and its related containment measures on the 341 mental health status of the general population across the lifespan. Moreover, the findings will 342 contribute to the further adaption of the self-help CBT programs. 343 In line with previous research findings, it is possible to predict that dropout rates may be higher with 344 web-based interventions than in traditional face-to-face therapy (80), especially when self-help 345 programs are used. To overcome this problem, participants in the study will receive a weekly 346 reminder and motivational messages to access the online material. A positive relationship between 347 each respondent and their referral therapist will be also supported, and while on the one hand, the 348 professional remains available in case of need, the subject takes responsibility over the course of the treatment. The learning process is emphasized, so to help the person improve self-management skillsand strategies to deal with their emotional problems.

Furthermore, the online format brings with it the advantage of allowing us to also support the population of Italians abroad, of which the literature does not report any in-depth analysis. RinascMENTE, therefore, represents the first attempt to provide online psychological support to the segment of the Italian population abroad.

## **CONCLUSION**

Since the beginning of the COVID-19 pandemic, studies demonstrated a significant clinical and statistically decrease in mental health across populations worldwide. This burden is expected to continue in the aftermath making high demand for timely and pragmatic psychological interventions tailored to the unique and immediate needs of the general public. Preventive measures, fear of being infected, and financial losses give a reason for the implementation and use of digital self-help programs based on CBT principles and techniques – which might offer a range of self-management strategies to cope with emotional difficulties, besides reducing the cost of the health care system (81).

# **DECLARATION**

## Ethics approval and consent to participate

The study protocol and informed consent to participate were approved by the Research Ethics Committee of the Catholic University of Milan, Italy (25-21). All participants will sign in the online informed consent to participate before entering the study.

## Consent for publication

Participants will give their consent for the anonymous publication of their data by signing the online informed consent form and information sheets

| 373 | Availability of data and materials |
|---|---|
| 374 | All data will be identified only by a code, with personal details kept in a secure online platform with |
| 375 | access only by the immediate research team. |
| 376 | |
| 377 | Competing interests |
| 378 | The authors declare that they have no competing interests. |
| 379 | |
| 380 | Funding |
| 381 | The author(s) received no financial support for the research, authorship, and/or publication of this |
| 382 | article. |
| 383 | |
| 384 | Authors' contributions |
| 385 | Conceptualization, V.B, M.S., and G.P.; methodology, G.P., and G.A.; writing—original draft |
| 386 | preparation, V.B., and M.S.; writing—review and editing, G.P., G.A., GMM, and G.C.; visualization |
| 387 | and supervision, G.P. and G.A.; project administration, G.P., and E.M. All authors have read and |
| 388 | agreed to the published version of the manuscript. |
| 389 | |
| 390 | Authors' contributions |
| 391 | Not applicable |
| 392 | |
| 393 | Trial status |
| 394 | Protocol Version 01 of February 2022 |
| 395 | Start of recruitment: 21/02/2022 |
| 396 | |
| 397 | REFERENCES |
| 398 | |

- 399 1. Bonaccorsi G, Pierri F, Cinelli M, Flori A, Galeazzi A, Porcelli F, et al. Economic and social
- 400 consequences of human mobility restrictions under COVID-19. Proceedings of the National
- 401 Academy of Sciences. 2020;117(27):15530-5.
- 402 2. Pietrabissa G, Volpi C, Bottacchi M, Bertuzzi V, Guerrini Usubini A, Loffler-Stastka H, et al.
- The Impact of Social Isolation during the COVID-19 Pandemic on Physical and Mental
- Health: The Lived Experience of Adolescents with Obesity and Their Caregivers.
- International journal of environmental research and public health. 2021;18(6).
- 406 3. Xiong J, Lipsitz O, Nasri F, Lui LMW, Gill H, Phan L, et al. Impact of COVID-19 pandemic
- on mental health in the general population: A systematic review. Journal of Affected
- 408 Disorders. 2020;277:55-64.
- 409 4. Nguyen HC, Nguyen MH, Do BN, Tran CQ, Nguyen TTP, Pham KM, et al. People with
- Suspected COVID-19 Symptoms Were More Likely Depressed and Had Lower Health-
- Related Quality of Life: The Potential Benefit of Health Literacy. Journal of Clinical
- 412 Medicine. 2020;9(4).
- 413 5. Rogers JP, Chesney E, Oliver D, Pollak TA, McGuire P, Fusar-Poli P, et al. Psychiatric and
- 414 neuropsychiatric presentations associated with severe coronavirus infections: a systematic
- review and meta-analysis with comparison to the COVID-19 pandemic. The lancet
- 416 Psychiatry. 2020;7(7):611-27.
- 417 6. Rajkumar RP. COVID-19 and mental health: A review of the existing literature. Asian Journal
- 418 of Psychiatry. 2020;52:102066.
- 7. Parola A, Rossi A, Tessitore F, Troisi G, Mannarini S. Mental Health Through the COVID-
- 420 19 Quarantine: A Growth Curve Analysis on Italian Young Adults. Frontiers in Psychology.
- 421 2020;11:567484.
- 422 8. Guerrini Usubini A, Cattivelli R, Varallo G, Castelnuovo G, Molinari E, Giusti EM, et al. The
- Relationship between Psychological Distress during the Second Wave Lockdown of COVID-

- 424 19 and Emotional Eating in Italian Young Adults: The Mediating Role of Emotional
- Dysregulation. Journal of personalized medicine. 2021;11(6).
- 426 9. Loffler-Stastka H, Bednar K, Pleschberger I, Prevendar T, Pietrabissa G. How to Include
- Patients' Perspectives in the Study of the Mind: A Review of Studies on Depression. Front
- 428 Psychol. 2021;12:651423.
- 429 10. Cao W, Fang Z, Hou G, Han M, Xu X, Dong J, et al. The psychological impact of the COVID-
- 430 19 epidemic on college students in China. Psychiatry Research. 2020;287:112934.
- 431 11. Pietrabissa G, Simpson SG. Psychological Consequences of Social Isolation During COVID-
- 432 19 Outbreak. Frontiers in psychology. 2020;11:2201.
- 433 12. Giusti EM, Pedroli E, D'Aniello GE, Stramba Badiale C, Pietrabissa G, Manna C, et al. The
- Psychological Impact of the COVID-19 Outbreak on Health Professionals: A Cross-Sectional
- Study. Frontiers in psychology. 2020;11:1684.
- 436 13. Ministero della Salute. Covid-19 Situazione nel mondo. 2021.
- 437 14. Bertuzzi V, Semonella M, Bruno D, Manna C, Edbrook-Childs J, Giusti EM, et al.
- 438 Psychological Support Interventions for Healthcare Providers and Informal Caregivers during
- the COVID-19 Pandemic: A Systematic Review of the Literature. International Journal of
- Environmental Research and Public Health. 2021;18(13).
- 441 15. Rossi Ferrario S, Panzeri A, Cerutti P, Sacco D. The Psychological Experience and
- Intervention in Post-Acute COVID-19 Inpatients. Neuropsychiatric disease and treatment.
- 443 2021;17:413-22.
- 444 16. Pietrabissa G, Manzoni GM, Algeri D, Mazzucchelli L, Carella A, Pagnini F, et al. Facebook
- 445 Use as Access Facilitator for Consulting Psychology. Australian Psychologist.
- 446 2015;40(4):299-303.
- 447 17. Rossi AA, Marconi M, Taccini F, Verusio C, Mannarini S. From Fear to Hopelessness: The
- Buffering Effect of Patient-Centered Communication in a Sample of Oncological Patients
- during COVID-19. Behav Sci (Basel). 2021;11(6).

- 450 18. Panzeri A, Rossi Ferrario S, Cerutti P. Psychological Differences Among Healthcare Workers
- of a Rehabilitation Institute During the COVID-19 Pandemic: A Two-Step Study. Frontiers
- in Psychology. 2021;12.
- 453 19. Maunder RG. Was SARS a mental health catastrophe? Gen Hosp Psychiatry. 2009;31(4):316–
- 454 7.
- 455 20. Schwartz R, Sinskey JL, Anand U, Margolis RD. Addressing Postpandemic Clinician Mental
- Health: A Narrative Review and Conceptual Framework. Annals of internal medicine.
- 457 2020;173(12):981-8.
- 458 21. Panzeri A, Rossi Ferrario S, editors. Supporting rehabilitation patients with COVID-19 during
- the pandemic: Experiences from a technology-based psychological approach. CEUR
- Workshop Proceedings: Second Symposium on Psychology-Based Technologies Psychobit,
- 461 2730; 2020.
- 462 22. Murphy R, Calugi S, Cooper Z, Dalle Grave R. Challenges and opportunities for enhanced
- cognitive behaviour therapy (CBT-E) in light of COVID-19. The Cognitive Behaviour
- 464 Therapist. 2020;13.
- 465 23. Jassi A, Shahriyarmolki K, Taylor T, Peile L, Challacombe F, Clark B, et al. OCD and
- 466 COVID-19: a new frontier. The Cognitive Behaviour Therapist. 2020;13.
- 467 24. Murray H, Grey N, Wild J, Warnock-Parkes E, Kerr A, Clark DM, et al. Cognitive therapy
- for post-traumatic stress disorder following critical illness and intensive care unit admission.
- The Cognitive Behaviour Therapist. 2020;13.
- 470 25. Wang C, Pan R, Wan X, Tan Y, Xu L, Ho CS, et al. Immediate Psychological Responses and
- Associated Factors during the Initial Stage of the 2019 Coronavirus Disease (COVID-19)
- Epidemic among the General Population in China. International journal of environmental
- 473 research and public health. 2020;17(5).
- 474 26. Kang L, Li Y, Hu S, Chen M, Yang C, Yang BX, et al. The mental health of medical workers
- in Wuhan, China dealing with the 2019 novel coronavirus. Lancet Psychiatry. 2020;7(3).

- 476 27. Shangguan F, Quan X, Qian W, Zhou C, Zhang C, Zhang XY, et al. Prevalence and correlates
- of somatization in anxious individuals in a Chinese online crisis intervention during COVID-
- 478 19 epidemic. Journal of Affective Disorders. 2020;277:436-42.
- 479 28. Brog NA, Hegy JK, Berger T, Znoj H. An internet-based self-help intervention for people
- with psychological distress due to COVID-19: study protocol for a randomized controlled
- 481 trial. Trials. 2021;22(1):171.
- Wei N, Huang BC, Lu SJ, Hu JB, Zhou XY, Hu CC, et al. Efficacy of internet-based integrated
- intervention on depression and anxiety symptoms in patients with COVID-19. Journal of
- 484 Zhejiang University Science B. 2020;21(5):400-4.
- 485 30. Pizzoli SMF, Marzorati C, Mazzoni D, Pravettoni G. An Internet-Based Intervention to
- 486 Alleviate Stress During Social Isolation With Guided Relaxation and Meditation: Protocol for
- a Randomized Controlled Trial. JMIR research protocols. 2020;9(6):e19236.
- 488 31. Barak A, Hen L, Boniel-Nissim M, Shapira N. A Comprehensive Review and a Meta-Analysis
- of the Effectiveness of Internet-Based Psychotherapeutic Interventions. Journal of
- 490 Technology in Human Services. 2008;26(2-4):109-60.
- 491 32. Griffiths KM, Farrer L, Christensen H. The efficacy of internet interventions for depression
- and anxiety disorders: a review of randomised controlled trials. Medical Journal of Australia.
- 493 2010;192(11).
- 494 33. Andersson G. Internet interventions: Past, present and future. Internet Interventions.
- 495 2018;12:181-8.
- 496 34. Liu S, Yang L, Zhang C, Xiang YT, Liu Z, Hu S, et al. Online mental health services in China
- during the COVID-19 outbreak. The lancet Psychiatry. 2020;7(4):e17-e8.
- 498 35. Castelnuovo G, Pietrabissa G, Manzoni GM, Sicurello F, Zoppis I, Molinari E. Fighting the
- 499 COVID-19 pandemic using the technology-based second-line in Italy and Lombardy: The
- urgent need of home-based remote monitoring systems to avoid the collapse of the hospital-
- centred first line. Journal of global health. 2020;10(2):010371.

- 502 36. Simpson S, Richardson L, Pietrabissa G, Castelnuovo G, Reid C. Videotherapy and
- therapeutic alliance in the age of COVID-19. Clinical psychology & psychotherapy.
- 504 2021;28(2):409-21.
- 505 37. Shafran R, Clark DM, Fairburn CG, Arntz A, Barlow DH, Ehlers A, et al. Mind the gap:
- Improving the dissemination of CBT. Behaviour research and therapy. 2009;47(11):902-9.
- 507 38. Nobili RM, Gambazza S, Spada MS, Tutino AL, Bulfamante AM, Mariani A, et al. Remote
- support by multidisciplinary teams: A crucial means to cope with the psychological impact of
- the SARS-COV-2 pandemic on patients with cystic fibrosis and inflammatory bowel disease
- in Lombardia. International journal of clinical practice. 2021;75(7):e14220.
- 39. Wang H, Zhao Q, Mu W, Rodriguez M, Qian M, Berger T. The Effect of Shame on Patients
- With Social Anxiety Disorder in Internet-Based Cognitive Behavioral Therapy: Randomized
- 513 Controlled Trial. JMIR mental health. 2020;7(7):e15797.
- Nordgreen T, Havik OE, Ost LG, Furmark T, Carlbring P, Andersson G. Outcome predictors
- in guided and unguided self-help for social anxiety disorder. Behaviour research and therapy.
- 516 2012;50(1):13-21.
- 41. Andersson G, Paxling B, Roch-Norlund P, Ostman G, Norgren A, Almlov J, et al. Internet-
- based psychodynamic versus cognitive behavioral guided self-help for generalized anxiety
- disorder: a randomized controlled trial. Psychotherapy and Psychosomatics. 2012;81(6):344-
- 520 55.
- 521 42. Van't Hof E, Cuijpers P, Stein DJ. Self-help and Internet-guided interventions in depression
- and anxiety disorders: a systematic review of meta-analyses. CNS spectrums. 2009;14(2)
- 523 Suppl 3):34-40.
- 524 43. Ciuca AM, Berger T, Crisan LG, Miclea M. Internet-based treatment for panic disorder: A
- three-arm randomized controlled trial comparing guided (via real-time video sessions) with
- 526 unguided self-help treatment and a waitlist control. PAXPD study results. Journal of Anxiety
- 527 Disorders. 2018;56:43-55.

- 528 44. Holst A, Nejati S, Bjorkelund C, Eriksson MC, Hange D, Kivi M, et al. Patients' experiences
- of a computerised self-help program for treating depression a qualitative study of Internet
- mediated cognitive behavioural therapy in primary care. Scandinavian Journal of Primary
- 531 Health Care. 2017;35(1):46-53.
- Reins JA, Boss L, Lehr D, Berking M, Ebert DD. The more I got, the less I need? Efficacy of
- Internet-based guided self-help compared to online psychoeducation for major depressive
- disorder. Journal of Affective Disorders. 2019;246:695-705.
- 535 46. Vernmark K, Lenndin J, Bjarehed J, Carlsson M, Karlsson J, Oberg J, et al. Internet
- administered guided self-help versus individualized e-mail therapy: A randomized trial of two
- versions of CBT for major depression. Behaviour research and therapy. 2010;48(5):368-76.
- 538 47. Andersson E, Enander J, Andren P, Hedman E, Ljotsson B, Hursti T, et al. Internet-based
- cognitive behaviour therapy for obsessive-compulsive disorder: a randomized controlled trial.
- Psychological Medicine. 2012;42(10):2193-203.
- 541 48. Ye YY, Chen NK, Chen J, Liu J, Lin L, Liu YZ, et al. Internet-based cognitive-behavioural
- therapy for insomnia (ICBT-i): a meta-analysis of randomised controlled trials. BMJ Open.
- 543 2016;6(11):e010707.
- 544 49. Coull G, Morris PG. The clinical effectiveness of CBT-based guided self-help interventions
- for anxiety and depressive disorders: a systematic review. Psychological medicine.
- 546 2011;41(11):2239-52.
- 547 50. Balestrieri M, Carta MG, Leonetti S, Sebastiani G, Starace F, Bellantuono C. Recognition of
- depression and appropriateness of antidepressant treatment in Italian primary care. Social
- Psychiatry and Psychiatric Epidemiology. 2004;39(3):171-6.
- 550 51. Goldberg DP. The Detection of Psychiatric Illness by Questionnaire: Oxford University Press:
- 551 Oxford.; 1972.
- 552 52. American Psychiatric Association. Diagnostic and statistical manual of mental disorders (5th
- ed.). Washington, DC2013.

- 53. Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G\*Power 3.1:
- Tests for correlation and regression analyses. Behavior Research Methods. 2009;41(4):1149-
- 556 60.
- 557 54. Pietrabissa G, Castelnuovo G, Jackson JB, Rossi A, Manzoni GM, Gibson P. Brief Strategic
- Therapy for Bulimia Nervosa and Binge Eating Disorder: A Clinical and Research Protocol.
- Front Psychol. 2019;10:373.
- 560 55. Cattivelli R, Castelnuovo G, Musetti A, Varallo G, Spatola CAM, Riboni FV, et al.
- ACTonHEALTH study protocol: promoting psychological flexibility with activity tracker and
- mHealth tools to foster healthful lifestyle for obesity and other chronic health conditions.
- 563 Trials. 2018;19(1):659.
- 564 56. Cohen J. Statistical power analysis for the behavioral sciences. press A, editor. London2013.
- 565 57. Eid M, Gollwitzer M, Schmitt M. Statistik und forschungsmethoden2017.
- 566 58. Castelnuovo G, Manzoni GM, Villa V, Cesa GL, Pietrabissa G, Molinari E. The STRATOB
- study: design of a randomized controlled clinical trial of Cognitive Behavioral Therapy and
- Brief Strategic Therapy with telecare in patients with obesity and binge-eating disorder
- referred to residential nutritional rehabilitation. Trials. 2011;12:114.
- 570 59. Chiappelli M, Lo Coco G, Gullo S, Bensi L, Prestano C. The Outcome Questionnaire 45.2.
- Italian validation of an instrument for the assessment of psychological treatments.
- 572 Epidemiologia e Psichiatria Sociale. 2008;17(2):152-61.
- 573 60. Mondo M, Sechi C, Cabras C. Psychometric evaluation of three versions of the Italian
- Perceived Stress Scale. Current Psychology. 2019:1-9.
- 575 61. Balzarotti S, John OP, Gross JJ. An Italian Adaptation of the Emotion Regulation
- Questionnaire. European Journal of Psychological Assessment. 2010;26(1):61-7.
- 577 62. Bottesi G, Ghisi M, Altoè G, Conforti E, Melli G, Sica C. The Italian version of the Depression
- Anxiety Stress Scales-21: Factor structure and psychometric properties on community and
- clinical samples. Comprehensive Psychiatry. 2015;60:170-81.

- 580 63. Wang C, Tee M, Roy AE, Fardin MA, Srichokchatchawan W, Habib HA, et al. The impact
- of COVID-19 pandemic on physical and mental health of Asians: A study of seven middle-
- income countries in Asia. PloS one. 2021;16(2):e0246824.
- 583 64. Wang C, Tripp C, Sears SF, Xu L, Tan Y, Zhou D, et al. The impact of the COVID-19
- pandemic on physical and mental health in the two largest economies in the world: a
- comparison between the United States and China. Journal of behavioral medicine.
- 586 2021;44(6):741-59.
- 587 65. Wang C, Lopez-Nunez MI, Pan R, Wan X, Tan Y, Xu L, et al. The Impact of the COVID-19
- Pandemic on Physical and Mental Health in China and Spain: Cross-sectional Study. JMIR
- formative research. 2021;5(5):e27818.
- 590 66. Soraci P, Ferrari A, Abbiati FA, Del Fante E, De Pace R, Urso A, et al. Validation and
- Psychometric Evaluation of the Italian Version of the Fear of COVID-19 Scale. Int J Ment
- 592 Health Addict. 2020:1-10.
- 593 67. Sibilia L, Schwarzer R, Jerusalem M. talian Adaptation of the General Self-Efficacy Scale:
- Self-Efficacy Generalizzata 1995 [Available from: <a href="http://userpage.fu-">http://userpage.fu-</a>
- 595 <u>berlin.de/~health/italian.htm.</u>
- 596 68. De Girolamo G, Rucci P, Scocco P, Becchi A, Coppa F, D'Addario A, et al. Quality of life
- assessment: validation of the Italian version of the WHOQOL-Brief. Epidemiologia e
- 598 Psichiatria Sociale. 2000;9(1):45-55.
- 599 69. Brooke J. SUS: A "quick and dirty" usability scale. In: Jordan PW, Thomas B, Weerdmeester
- BA, McClelland IL, editors. Usability evaluation in industry. London: Taylor & Francis;
- 601 1996. p. 189-94.
- Vlaescu G, Alasjo A, Miloff A, Carlbring P, Andersson G. Features and functionality of the
- Iterapi platform for internet-based psychological treatment. Internet Interventions.
- 604 2016;6:107-14.

- 605 71. Semonella M, Vilchinsky N, Dakel R, Biliunaite I, Pietrabissa G, Andersson G, editors.
- SOSteniamoci: An internet-based intervention to support informal caregivers. PSYCHOBIT;
- 607 2020.
- Thoren ES, Oberg M, Wanstrom G, Andersson G, Lunner T. A randomized controlled trial
- evaluating the effects of online rehabilitative intervention for adult hearing-aid users.
- International journal of audiology. 2014;53(7):452-61.
- Hesser H, Gustafsson T, Lunden C, Henrikson O, Fattahi K, Johnsson E, et al. A randomized
- controlled trial of Internet-delivered cognitive behavior therapy and acceptance and
- commitment therapy in the treatment of tinnitus. Journal of consulting and clinical
- psychology. 2012;80(4):649-61.
- 74. Tulbure BT, Szentagotai A, David O, Stefan S, Mansson KN, David D, et al. Internet-
- delivered cognitive-behavioral therapy for social anxiety disorder in Romania: a randomized
- 617 controlled trial. PloS one. 2015;10(5):e0123997.
- 5. Johansson R, Sjoberg E, Sjogren M, Johnsson E, Carlbring P, Andersson T, et al. Tailored vs.
- standardized internet-based cognitive behavior therapy for depression and comorbid
- symptoms: a randomized controlled trial. PloS one. 2012;7(5):e36905.
- 621 76. IBM Corp. IBM SPSS Statistics for Windows, Version 24.0. In: Armonk NIC, editor.
- 622 Released 2016.
- 623 77. Barak A, Grohol JM. Current and future trends in internet-supported mental health
- interventions. Journal of Technologies at Human Services. 2011;29:155–96.
- Newman MG, Szkodny LE, Llera SJ, Przeworski A. A review of technology-assisted self-
- help and minimal contact therapies for anxiety and depression: is human contact necessary for
- therapeutic efficacy? Clinical psychology review. 2011;31(1):89-103.
- 628 79. Liverpool S, Mota CP, Sales CMD, Cus A, Carletto S, Hancheva C, et al. Engaging Children
- and Young People in Digital Mental Health Interventions: Systematic Review of Modes of
- Delivery, Facilitators, and Barriers. Journal of medical Internet research. 2020;22(6):e16317.

80. Botella C, Mira A, Herrero R, García-Palacios A, Baños R. Un programa de intervención autoaplicado a través de Internet para el tratamiento de la depresión: "Sonreír es divertido".
Aloma. 2015;33(2):39-48.
81. Castelnuovo G, Pietrabissa G, Cattivelli R, Manzoni GM, Molinari E. Not Only Clinical
Efficacy in Psychological Treatments: Clinical Psychology Must Promote Cost-Benefit, CostEffectiveness, and Cost-Utility Analysis. Front Psychol. 2016;7:563.